CLINICAL TRIAL: NCT06885190
Title: Multisensory Processing of Alcohol Cues in Young Adult Binge Drinkers
Status: Not yet recruiting | Type: Observational
Sponsor: Rochester Institute of Technology (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Rebecca Houston, Associate Professor, Rochester Institute of Technology
Other Study IDs: SRS00020124; R15AA031579-01A1 (NIH)
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Drinking, Binge
Keywords: alcohol; young adult; multisensory; cues; event-related potentials; virtual reality
MeSH Terms: conditions — Binge Drinking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Young Adult Binge Drinkers: Participants ages 18 to 25 with a history of binge drinking (at least 2 episodes of 5+ standard drinks per episode for males/4+ standard drinks per episode for females) in the past month and at least 4+/3+ (males/females) score on the Alcohol Use Disorder Identification Test.
- Young Adult Social Drinkers: Participants ages 18 to 25 who report drinking alcohol at least once in the past month but no current history of a binge pattern (i.e., 2 or fewer drinks per episode) AND score less than 4/3 (males/females) on the Alcohol Use Disorder Identification Test.

SUMMARY:
Binge drinking is common among young adults and is related to many negative health outcomes including blackouts, risky sex, drunk driving, alcohol use disorder, and liver disease. Understanding whether there are differences in how binge drinkers respond to alcohol-related cues and whether this is related to craving is important for improving interventions and treatments. The proposed study will compare behavioral and neural processing of alcohol and non-alcohol cues in a single sensory modality (vision) with that of cues presented in multiple sensory modalities (vision, touch, and smell) with varying degrees of realistic appearance (images, virtual reality, real objects). Participants will answer questionnaires related to their physical and mental health and recent alcohol and drug use. Those eligible for the study will complete two in-person lab sessions. During both sessions they will be asked to view a series of cues which will include images on a computer screen, objects presented in virtual reality, or real objects. Sometimes these will be presented just visually and other times they will be combined with the presentation of specific smells or an object to touch. Some of these cues will be alcohol-related and others will be neutral (non-alcohol-related). Brainwave activity, as measured by the electroencephalogram (EEG), and reports of alcohol craving will be collected during these sessions. It is expected that brainwave activity will be greatest in response to multisensory cues compared to that in response unisensory (visual only) cues. It is also expected that young adults with a recent history of binge drinking will show the greatest brainwave activity in response to multisensory alcohol cues compared to social drinkers. Binge drinkers will also report more alcohol craving in response to multisensory alcohol cues compared to social drinkers. It is anticipated that brainwave responses will increase as the level of realism of the cues increases. Binge drinkers will also show stronger brainwave and craving responses to multisensory alcohol cues presented as real objects. Finally, binge drinkers will show lessened brain and craving responses when multisensory cues do not match compared to social drinkers. For example, if a photo shows an alcoholic drink but the smell presented is not alcohol related, binge drinkers will show less attentive brain activity toward those mismatched cues. Given that most alcohol cues in daily life are experienced across multiple senses simultaneously, results of this research will provide a better understanding of the relation between alcohol cue processing and craving, and will inform development of more effective programs for decreasing young adult risky drinking behavior.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 to 25 years old
* meet criteria for either the binge drinker or social drinker groups previously described

Exclusion Criteria:

* history of head injury involving loss of consciousness of 10+ minutes
* colorblindness
* hearing, tactile, olfactory or uncorrected vision deficits
* history of seizures
* neurological disorder diagnosis
* mental health history of psychosis or mania
* history of alcohol or substance use disorder diagnosis
* illicit drug use in the past 30 days
* changes to psychotropic medication type or dose in past 3 months

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited via social media advertisements, fliers posted on college campuses and in the community, and a departmental research participants group.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Event-related Potential Amplitudes in Response to Alcohol and Neutral Cues | Baseline and follow-up (within 1 week)
  Amplitude (magnitude) of electrocortical activity assessed in response to alcohol-related and neutral cues presented either visually or in visual-olfactory or visual-tactile combinations.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Houston, PhD, Principal Investigator — Rochester Institute of Technology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill-Bowen LD, Riedel MC, Poudel R, Salo T, Flannery JS, Camilleri JA, Eickhoff SB, Laird AR, Sutherland MT. The cue-reactivity paradigm: An ensemble of networks driving attention and cognition when viewing drug and natural reward-related stimuli. Neurosci Biobehav Rev. 2021 Nov;130:201-213. doi: 10.1016/j.neubiorev.2021.08.010. Epub 2021 Aug 13. PMID 34400176
- [Background] Connor JP, Kavanagh DJ, Andrade J, May J, Feeney GF, Gullo MJ, White AM, Fry ML, Drennan J, Previte J, Tjondronegoro D. Alcohol consumption in young adults: the role of multisensory imagery. Addict Behav. 2014 Mar;39(3):721-4. doi: 10.1016/j.addbeh.2013.11.023. Epub 2013 Dec 4. PMID 24360399
- [Background] Kiyak C, Simonetti ME, Norton S, Deluca P. The efficacy of cue exposure therapy on alcohol use disorders: A quantitative meta-analysis and systematic review. Addict Behav. 2023 Apr;139:107578. doi: 10.1016/j.addbeh.2022.107578. Epub 2022 Dec 12. PMID 36563480
- [Background] Mellentin AI, Skot L, Nielsen B, Schippers GM, Nielsen AS, Stenager E, Juhl C. Cue exposure therapy for the treatment of alcohol use disorders: A meta-analytic review. Clin Psychol Rev. 2017 Nov;57:195-207. doi: 10.1016/j.cpr.2017.07.006. Epub 2017 Jul 27. PMID 28781153
- [Background] Hone-Blanchet A, Wensing T, Fecteau S. The use of virtual reality in craving assessment and cue-exposure therapy in substance use disorders. Front Hum Neurosci. 2014 Oct 17;8:844. doi: 10.3389/fnhum.2014.00844. eCollection 2014. PMID 25368571